CLINICAL TRIAL: NCT04146012
Title: Bovine Early Access, Compatibility and Hemostasis Post-Market Trial to Evaluate the Safety and Effectiveness of Early Access in Patients Who Require an Arteriovenous Conduit for Hemodialysis Using the Artegraft® Collagen Vascular Graft™
Brief Title: BEACH Trial: Bovine Early Access, Compatibility and Hemostasis Trial
Acronym: BEACH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company was sold and clinical trial was suspended then teminated
Sponsor: Artegraft, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARTCT.BEACH.001
Record Dates: First submitted 2019-10-21; First posted 2019-10-31 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Renal Insufficiency,Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Artegraft will follow all study patients enrolled in the proposed clinical trial and that have successful cannulation within 72 hours as defined above, for 6 months. If follow-up is necessary at 1 year after graft implantation, it will be done via phone survey. The late-access group [>/= 10 days] will be followed to 30 days post-first cannulation. If follow-up is necessary at 6 months after graft implantation, it will be done via phone survey. Day 0 is defined as the day of first cannulation, for early-access and late-access groups, to allow full follow-up to at least 30 days for both groups.
Who Masked: Investigator
Masking Description: Patients will be randomized in a 2:1 ratio to either early or late vascular access. The randomization will be stratified by investigative site, and will use a random permuted block design within strata, with blocks of size 3 and 6 ordered randomly within site.
  Once a patient signs informed consent, is determined to meet the inclusion/exclusion criteria, and is successfully implanted with the Artegraft, the site designated staff will open an envelope to determine the randomization number and whether the patient is randomly allocated to early or late vascular access.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Early Access (Active Comparator): Artegraft® Collagen Vascular Graft™ (Artegraft) will be accessed in less than 72 hours after implantation.
  Interventions: Device: Artegraft® Collagen Vascular Graft™ (Artegraft)
- Normal Access (Active Comparator): Artegraft® Collagen Vascular Graft™ (Artegraft) will be accessed after 10 days as per current IFU.
  Interventions: Device: Artegraft® Collagen Vascular Graft™ (Artegraft)

INTERVENTIONS:
Device: Artegraft® Collagen Vascular Graft™ (Artegraft) — The Artegraft is intended for use distal to the aorta as a segmental arterial replacement, as an arterial bypass, as an arteriovenous shunt where more conventional methods have proven inadequate, or as an arterial patch graft.

SUMMARY:
Bovine Early Access, Compatibility, and Hemostasis (BEACH) Trial Study is to evaluate the Safety and Effectiveness of Early Access in Patients Who Require an Arteriovenous Conduit for Hemodialysis using the Artegraft® Collagen Vascular Graft™. The objective of the BEACH Trial is to demonstrate that early access of Artegraft is associated with acceptable rates of successful early access, and acceptable rates of a composite of adverse events, to support a modification of existing device labeling stating that Artegraft is capable of cannulation within 72 hours post implantation.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major health problem that affects approximately 26 million Americans. Many of those suffering CKD will progress to develop end stage renal disease (ESRD) and require lifelong hemodialysis (HD) to filter wastes from their blood. There are nearly 2.5 million patients who receive HD worldwide, and this population is growing at a rate of 8% per year. This projects that the worldwide HD population to reach approximately 3.4 million by the year 2020. There are over 600,000 patients on HD in the US and an estimated 100,000 new cases are reported annually. The interventions required to maintain a person on HD carry a significant financial burden, with costs estimated to be as high as $30 billion annually. Given the increasing epidemic of obesity, diabetes, and heart disease, the burden of ESRD will continue to grow, making new interventions that can improve the social, physical, and financial realities of treating ESRD essential.

A critical factor in the survival of renal dialysis patients is the surgical creation of vascular access. Despite the fistula-first initiative, many patients will start hemodialysis using a central venous catheter (CVC). This increases the risks of associated bloodstream infections, central venous stenosis, and poorer outcomes from subsequent vascular cannulations.

Arteriovenous grafts have advantages compared with central venous catheters for dialysis and guidelines suggest their use as second choice after arteriovenous fistulas. The suggested advantages of grafts over fistulas is the ability to cannulate or access the graft earlier, traditionally 2 weeks for AVG rather than 6 weeks for AVF, and the lower rates of primary failure.

Standard practice with expanded polytetrafluoroethylene (ePTFE) grafts has been to avoid cannulation for 2 weeks following placement, but new generation grafts have been marketed for their early cannulation properties allowing use as an alternative to central venous catheters for prompt access.

The proposed BEACH Trial is a multi-center, prospective clinical trial to evaluate early access of an existing, FDA-approved bovine carotid vascular graft, approved as a general peripheral vascular graft and for hemodialysis. The BEACH Trial is seeking to demonstrate that early access, defined as within 72 hours post implantation, of the Artegraft device results in acceptable clinical outcomes including ability to support dialysis needs thereby obviating the requirement for interim catheter placement or facilitating the removal of an existing catheter with acceptable composite major adverse clinical events (MACE) rate up to 26 weeks (6 months) post implant.

Few vascular products approved in the 1970s have a broad level of acceptance in today's competitive market. Review of the original NDA application for Artegraft as well as the scientific literature revealed no clinical rationale for a waiting period of 14 days (for most access grafts) and 10 days (for Artegraft) before cannulation. The current literature does not seem to support the current guidelines as there is no evidence to suggest that a delay in cannulation of PTFE grafts will improve graft survival and patency.Note also that Artegraft cannot identify any scientific justification in the original NDA for the warning that was placed in the IFU to support the 10-day waiting period before cannulation.

Further, if it is assumed that dialysis is conducted 3 times per week, by allowing cannulation to the Artegraft device in the 72-hour period, only 6 to 10 additional needle punctures are added during the first 10-day period depending on whether cannulation is initiated within 72 hours, respectively. Artegraft believes that this limited number of additional early needle punctures will not significantly affect the safety or efficacy of the graft or the cannulation procedure.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet the following criteria:

1. Male or Female, 18 years or older
2. Diagnosis of End Stage Renal Disease (ESRD) and require vascular access for hemodialysis
3. Native [autogenous tissue] AV fistula creation or access is not indicated or non-viable [disadvantaged veins]
4. Requiring repair of an existing fistula or conduit, but only if using Artegraft as an interposition placement and the Artegraft is cannulated [not the fistula]. Artegraft must be place in a fresh subcutaneous tunnel. Thigh loop grafts will not be used.
5. Able to accommodate vascular graft placement in the upper extremity (i.e., forearm, or upper arm)
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF)
7. Able and willing to comply with the study protocol
8. Agrees to initiate and maintain hemodialysis treatments
9. Life expectancy is > 1 year based on physician assessment

Exclusion Criteria:

Patients are excluded from the trial if any of the following criteria apply:

1. High grade central venous stenosis/occlusion
2. Breast-feeding, pregnant or planning pregnancy within next 12 months.
3. Non-resolved infected existing grafts
4. Documented sepsis/bacteremia by blood culture within 4 weeks of implantation.
5. History of non-controlled immunodeficiency syndrome, including AIDS/HIV; Active clinically significant immune-mediated disease, not controlled by low-dose maintenance immunosuppression. The diagnosis of HIV alone, provided adequately treated, is not a contraindication for enrolment.
6. Severe liver dysfunction and/or coagulation or bleeding disorders.
7. Elevated platelet count > 1 million cells/mm3
8. History of heparin-induced thrombocytopenia syndrome (HIT)
9. Documented hypercoagulable state
10. Currently participating in another investigational drug or device study which may clinically interfere with any endpoints of this trial
11. Known hypersensitivity or contraindication to device materials or procedural medications that cannot be adequately managed medically
12. History or evidence of severe cardiac disease (NYHA Functional Class III or IV), , myocardial infarction within 6 months of enrollment, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina, uncontrolled CHF
13. History or evidence of severe peripheral arterial disease in the extremity selected for implant (i.e. arterial inflow insufficient to support hemodialysis)
14. History of cancer with active disease or treatment within the previous year, except for non-invasive basal or squamous cell carcinoma of the skin
15. Bleeding diathesis, other than that associated with ESRD
16. Scheduled renal transplant within 6 months
17. Patients who require chronic anticoagulation except for antiplatelet therapy. Patients currently receiving or who have received within the last month direct thrombin inhibitors, factor Xa inhibitors, or vitamin K antagonists should not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Malas, MD, Principal Investigator — University of California, San Diego
Locations (5):
- United States (5):
  - University of California, San Diego, California
  - Capital District Renal Physicians, Albany, New York
  - Dialysis Access Institute, Orangeburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - City Hospital at White Rock, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
No plans to share individual patient data

REFERENCES:
- [Background] Manns B, Tonelli M, Yilmaz S, Lee H, Laupland K, Klarenbach S, Radkevich V, Murphy B. Establishment and maintenance of vascular access in incident hemodialysis patients: a prospective cost analysis. J Am Soc Nephrol. 2005 Jan;16(1):201-9. doi: 10.1681/ASN.2004050355. Epub 2004 Nov 24. PMID 15563567
- [Background] Pastan S, Soucie JM, McClellan WM. Vascular access and increased risk of death among hemodialysis patients. Kidney Int. 2002 Aug;62(2):620-6. doi: 10.1046/j.1523-1755.2002.00460.x. PMID 12110026
- [Background] Al Shakarchi J, Inston N. Timing of cannulation of arteriovenous grafts: are we too cautious? Clin Kidney J. 2015 Jun;8(3):290-2. doi: 10.1093/ckj/sfu146. Epub 2015 Jan 20. PMID 26034590
- [Background] US Renal Data System, Annual Data Report: Atlas of Chronic Kidney Disease and End Stage Renal Disease in the United States, Bethesda MD, National Institutes of Health, National Institute of Diabetes and Kidney Diseases, 2009
- [Background] Fresenius Medical Care : Fresenious Medical Care Annual Report 2011 - Dialysis Market, Bad Homburg, Germany, Freesenious Medical Care, 2011
- [Background] US Renal Data System: 2012 Annual Data Report : Atlas of Chronic Kidney Disease and End-Stage Renal Disease in the United States, Bethesda, MD, National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, 2012
- [Background] US Renal Data System: 2014 Annual Data Report : Atlas of Chronic Kidney Disease and End-Stage Renal Disease in the United States, Bethesda, MD, National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, 2014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated (Sale of Company) First patient implanted 3 Dec 2019 Last Patient implanted 16 Dec 2019
Period: Overall Study
Arm/Group | Early Access | Normal Access
Started | 33 | 17
Completed | 3 | 2
Not Completed | 30 | 15
Not completed — Study Terminated | 30 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Access | Normal Access | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Successfully Cannulated.
Description: Early access success, defined by three cannulations, the first one started within 72 hours after implantation, all with minimum dialysis flow rates of 250 ml/min pump flow rate, with a minimum 17-gauge needle.
Time Frame: less than 72 hours
Population: No statistical analysis of data was conducted.
Measure: Number; unit: participants
Arm/Group | Early Access | Normal Access
Number analyzed (Participants) | 3 | 2
participants | 3 | 2

2. Primary Outcome: Patients That Experienced Major Adverse Events
Description: A composite of major adverse clinical events (MACE) including perigraft infection, hemorrhage / hematoma, thrombosis, and pseudoaneurysm within 30 days after first cannulation [Day 0] in the early-access and late-access groups.
Time Frame: Less than 6 month
Population: No statistical analysis of data was conducted.
Measure: Number; unit: Events
Arm/Group | Early Access | Normal Access
Number analyzed (Participants) | 3 | 2
Events | 0 | 0

3. Secondary Outcome: Grafts That Were Patent After 30 Days
Description: Patency (Primary, Assisted Primary, and Secondary) at 30 days after first successful cannulation [Day 0], and at 12 and 6 months after implantation in the early-access group and at 30 days post-Day 0 in the late-access group. The late access group will also be assessed for patency at 6 months through a telephone interview or office visit to provide a more robust data set.
Time Frame: Less than 6 months
Population: No statistical analysis of data was conducted..
Measure: Count of Participants; unit: Participants
Arm/Group | Early Access | Normal Access
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

4. Secondary Outcome: Patients That Experience Major Adverse Events
Description: All adverse events will be collected in the early-access group [to 6 months] and the late-access group [to 30 days post Day 0] and summarized by unique event, seriousness, and relationship to device or procedure.
Time Frame: Less than 6 months
Population: No statistical analysis of data was conducted.
Measure: Number; unit: Events
Arm/Group | Early Access | Normal Access
Number analyzed (Participants) | 3 | 2
Events | 0 | 0

5. Secondary Outcome: Removal of Catheter After Implantation (For Information Only)
Description: The number of days from graft implant or fistula revision to catheter removal shall be recorded.
Time Frame: Less than 6 months
Population: Data was not collected
Arm/Group | Early Access | Normal Access
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data was collect over 26 week period
Arm/Group | Early Access | Normal Access
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT04146012/Prot_SAP_000.pdf